CLINICAL TRIAL: NCT03729726
Title: A Randomized Controlled Trial Study of the Future Foundation 2.0 Personal Responsibility Education Innovative Strategies (PREIS) Program
Brief Title: Future Foundation 2.0 Personal Responsibility Education Innovative Strategies (PREIS) Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Metis Associates, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Future Foundation, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MetisIRBFFPREIS05062017
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Teen Pregnancy; Pregnancy in Adolescence; Teen Pregnancy Prevention; Pregnancy Prevention; Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Future Foundation 2.0 PREIS Program (Experimental): The Future Foundation 2.0 PREIS intervention model will include: a mandatory school-year program that offers after-school programming 4 days a week, including 120 hours of education (direct instruction & homework support), 30 hours of health (social emotional learning & sexual health), and 15 hours of student advocacy; an optional, 4-week summer program that offers 120 hours of programming each summer, including 16 hours of health (social emotional learning - service learning), 104 hours of project-based learning and enrichment (project-based learning in STEM - 64 hours) and enrichment (i.e., field trips, career speakers, and arts and crafts opportunities- 40 hours); and an optional parent engagement program, which will offer monthly parent workshops and quarterly events.
  Interventions: Behavioral: Future Foundation 2.0 PREIS Program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Future Foundation 2.0 PREIS Program — The Future Foundation 2.0 PREIS intervention model uses a placed-based collective impact framework to provide a comprehensive intervention model, including: academic support and college and career readiness services, evidence-based social emotional learning instruction to strengthen protective factors and promote healthy transitions to adulthood, and trauma-informed, medically accurate, and age appropriate sexual health education. Moreover, the 2.0 PREIS program model features a unique student advocacy component designed to ensure that youth and their families receive the wraparound supports necessary for their students to remain on track for school success.
  Arms: Future Foundation 2.0 PREIS Program

SUMMARY:
This study uses a randomized controlled trial (RCT) design to evaluate the impacts of the Future Foundation (FF) 2.0 Personal Responsibility Education Innovative Strategies (PREIS) program on reducing students' sexual activity (vaginal), recent risking sexual activity without condom use, and unprotected sex (no condoms/contraceptives). FF will implement the 2.0 PREIS Program with three cohorts of African-American youth in the 6th to 8th grades. FF aims to recruit and enroll 400 students who are new to the program for Cohort 1, 150 new students for Cohort 2, and another 150 new students for Cohort 3. These cohorts of eligible students will come from grades 6-8 in Woodland and McNair middle schools and projected to attend Banneker high school. Random assignment will be an ongoing process throughout the project enrollment periods. By the end of the recruitment processes, a total of 700 students will be randomly assigned to either the treatment or the control group, resulting in 350 students in each condition. Each year, the FF 2.0 PREIS intervention model will offer year-round grant-funded services, including after-school, summer programming, and parent engagement activities. The 350 youth randomly assigned to the treatment group will be offered the FF 2.0 PREIS program (Cohort 1 will target 200 treatment youth from January 2018 through June 2018; Cohort 2 will target 75 treatment youth from August 2018 through May 2019; and Cohort 3 will serve 75 treatment youth from August 2019 through May 2020.), while the 350 students assigned to the control group may receive after school and/or summer programming from another community-based organization. The primary hypotheses for the RCT study are the following: significantly fewer numbers of students in the FF 2.0 PREIS intervention engage in vaginal sex than their control group peers do by the time of the end of the program and also at the six-month follow-up; significantly fewer numbers of students in the FF 2.0 PREIS intervention engage in recent unprotected sex significantly than the control group students do at the end of the program and also at the six-month follow-up; and significantly greater numbers of participants in the FF 2.0 PREIS intervention remain abstinent or report condom use during recent vaginal sexual activity than the control group students do at the end of the program and also at the six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Schools: attending Woodland and McNair middle schools and projected to attend Banneker high school
* Grade level: Grades 6-8
* Race/ethnicity or tribe: 100% African American
* Gender: 34% male and 66% female (based on current make-up of Future Foundation youth)
* Risk characteristics: 93% of youth will come from low-income families (based on free lunch eligibility)
* Other characteristics: The majority of target youth will also exhibit academic need. 81% will be below proficiency in English language arts and 90% will score not proficient in math. All recruited subjects will be new to Future Foundation services.

Exclusion Criteria:

* Students who have already received Future Foundation services

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Post measure of ever having vaginal sex in the past 3 months | 12 months after baseline
  A dichotomous measure collected at the end of the program based on self-report questionnaire.
Post measure of risk of exposure to sexually transmitted infections in the past 3 months | 12 months after baseline
  A dichotomous measure collected at the end of the program based on self-report questionnaire.
Post measure of ever having unprotected vaginal sex in the past 3 months | 12 months after baseline
  A dichotomous measure collected at the end of the program based on self-report questionnaire.
Follow-up measure of ever having vaginal sex in the past 3 months | 18 months after baseline
  A dichotomous measure collected six months after the end of program implementation based on self-report questionnaire.
Follow up measure of risk of exposure to sexually transmitted infections in the past 3 months | 18 months after baseline
  A dichotomous measure collected six months after the end of program implementation based on self-report questionnaire.
Follow up measure of ever having unprotected vaginal sex in the past 3 months | 18 months after baseline
  A dichotomous measure collected six months after the end of program implementation based on self-report questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Future Foundation, East Point, Georgia, United States